CLINICAL TRIAL: NCT03687970
Title: A New Method for Identifying Sensory Changes in Painful Chemotherapy-induced Peripheral Neuropathy (CIPN): a Feasibility Study
Brief Title: A New Method for Identifying Sensory Changes in Painful Chemotherapy-induced Peripheral Neuropathy (CIPN)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Lasmed LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 201807162; 1R43CA206796-01A1 (NIH)
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Results first posted 2020-10-22 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: CIPN; Neuropathic pain; DLss; Peripheral neuropathy
MeSH Terms: conditions — Neuralgia; Peripheral Nervous System Diseases | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Painful CIPN Group (Experimental): -Performed at baseline: NPSI, BPI, HADS, Spontaneous pain at baseline on 0-10 Numerical Rating Scale (NRS), QST, CPM, and DLss
  Interventions: Other: Brief Pain Inventory; Other: Hospital Anxiety and Depression Scale; Other: Neuropathic Pain Symptom Inventory; Procedure: Diode Laser fiber type Selective Stimulator; Procedure: Quantitative sensory testing; Procedure: Conditioned pain modulation efficiency; Other: Spontaneous pain at baseline on 0-10 Numerical Rating Scale (NRS)
- Group B: Control Group (Active Comparator): -Performed at baseline: NPSI, BPI, HADS, Spontaneous pain at baseline on 0-10 Numerical Rating Scale (NRS), QST, CPM, and DLss
  Interventions: Other: Brief Pain Inventory; Other: Hospital Anxiety and Depression Scale; Other: Neuropathic Pain Symptom Inventory; Procedure: Diode Laser fiber type Selective Stimulator; Procedure: Quantitative sensory testing; Procedure: Conditioned pain modulation efficiency; Other: Spontaneous pain at baseline on 0-10 Numerical Rating Scale (NRS)

INTERVENTIONS:
Other: Brief Pain Inventory — -A self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. The patient is asked to rate their worst, least, average, and current pain intensity (4 items which generate the PAIN SEVERITY score), list current treatments and their perceived effectiveness, and rate the degree that pain interferes with general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life (7 items which generate the PAIN INTERFERENCE score) on a 10 point scale.
  Other Names: BPI
Other: Hospital Anxiety and Depression Scale — * 14 item scale with even of the items relating to anxiety and seven relating to depression
  * Each item on the questionnaire is scored from 0-3 and this means that a patient can score between 0 and 21 for either anxiety or depression
  Other Names: HADS
Other: Neuropathic Pain Symptom Inventory — -The NPSI questionnaire utilized in this study includes eight parameters (i.e., burning pain, squeezing pain, pressure pain, electric shock pain, stabbing pain, tingling pain, pins and needles pain and allodynia [pain provoked by light touch]). Each of the parameters includes recall of the past 24 hours
  Other Names: NPSI
Procedure: Diode Laser fiber type Selective Stimulator — -Each patient will have an A and C fiber stimulation. Stimulation will be performed on the dorsum of the foot using stimulation previously published parameters to elicit "burning pain," which is from activation of C-fibers and "pinprick" pain from A-fibers
  Other Names: DLss
Procedure: Quantitative sensory testing — * Quantitative sensory testing will be performed on the dorsal mid-foot and the ipsilateral shoulder will serve as control area
  * Cold and warm detection thresholds, cold and heat pain thresholds, mechanical detection thresholds, and wind-up ratio
  Other Names: QST
Procedure: Conditioned pain modulation efficiency — -Immersion of a hand up to the wrist to a thermostat-controlled water bath maintained at 12 degrees Celsius, and the application of a heat stimulus on the contralateral forearm.
  Other Names: CPM
Other: Spontaneous pain at baseline on 0-10 Numerical Rating Scale (NRS) — -The subjects are asked to rate the intensity of their current pain on a 0-10 scale - 0 denoting "no pain" and 10 denoting "worst imaginable pain".

SUMMARY:
The investigators propose that using the Diode Laser fiber type Selective Stimulator (DLss) in patients with chemotherapy-induced peripheral neuropathy (CIPN) will allow for the assessment of changes in small-fiber pain thresholds, to identify differences between subjects who received chemotherapy and developed painful CIPN, compared to subjects who received similar chemotherapy but did not develop painful CIPN (control group).

Additionally, the investigators would like to investigate whether the response to DLss correlates with pain severity in patients with persistent painful neuropathy.

The ultimate goal of this study is to develop a non-invasive, bedside quantitative test that is specific for painful CIPN. If the investigators' initial hypothesis is confirmed, the next step would be to design a prospective longitudinal study and assess changes in DLss early after initiation of chemotherapy, to determine whether this approach can help identify early predictive parameters of painful CIPN.

DETAILED DESCRIPTION:
Painful chemotherapy-induced peripheral neuropathy (CIPN) is a common side effect of chemotherapy, occurring in more than 60% of patients at some point during the course of cancer treatment with commonly used drugs such as taxanes and platinum compounds. It potentially may result in severely diminished quality of life and dose reduction or/and treatment delay, which may ultimately impact survival.

The mechanisms by which chemotherapy-induced nerve damage ultimately leads to pain are poorly understood, because virtually no structural or functional differences in nerve fibers between painless and painful peripheral neuropathy have been identified. As a result, there is no reliable way to predict which patients will develop persistent painful chemotherapy-induced peripheral neuropathy.

The ultimate goal of this study is to develop a non-invasive, bedside quantitative test that is specific for painful CIPN. If our initial hypothesis is confirmed, the next step would be to design a prospective longitudinal study and assess changes in DLss early after initiation of chemotherapy, to determine whether this approach can help identify early predictive parameters of painful CIPN.

In this other interventional study, we will test the utility of the Diode Laser fiber type Selective Stimulator (DLss) to identify sensory changes that are unique to patients with painful chemotherapy induced peripheral neuropathy (CIPN) vs. controls.

Painful symptoms of CIPN develop in patients with differential nerve damage to Aδ vs C-type peripheral nerve fibers. We hypothesize that Aδ:C fiber threshold ratio, as measured by the DLss, will be different between patients with painful CIPN compared to control patients who received a similar regimen of chemotherapy, but did not develop painful CIPN. The confirmation of hypothesis may lead to a novel approach for early detection of CIPN.

Subjects: 20 evaluable patients with painful CIPN following treatment with oxaliplatin, cisplatin, paclitaxel, docetaxel (or any combination of above) will be included in painful CIPN group, and 20 controls matched by the type of chemotherapy received, who did not develop painful CIPN.

The study procedure will include a one-time visit for sensory assessments including:

1. Spontaneous pain at baseline on 0-10 Numerical Rating Scale (NRS);
2. Assessment of pain symptoms on Neuropathic pain Symptom Inventory (NPSI) and Brief Pain Inventory (BPI).
3. Assessment of mood on hospital anxiety and depression scale (HADS)
4. Quantitative sensory testing (QST): thermal detection and pain thresholds, mechanical detection threshold, temporal summation (TS), and conditioned pain modulation (CPM).

The primary outcome is the comparison of Aδ:C fiber threshold ratio between patients who have developed painful CIPN, and the control subjects.

In secondary analyses, we will generate Spearman correlation coefficient between the "Aδ:C fiber threshold ratio" and the severity of painful CIPN on NPSI scale.

ELIGIBILITY:
Inclusion Criteria:

Group A: Painful CIPN group

* Age >18
* Distal symmetric pain distribution (both feet, with or without pain in hands).
* The pain appeared during or up to 12 weeks after treatment with oxaliplatin, cisplatin, paclitaxel, docetaxel or any combination of these.
* Score of 4 or more on Douleur Neuropathique 4 (DN4) neuropathic pain questionnaire
* Pain duration > 2 months.
* Patient report of average daily pain intensity in the last week ≥3 on 0-10 Numerical Rating Scale (NRS).
* Able and willing to sign an Institutional Review Board (IRB)-approved written informed consent.

Group B: Control group:

* Age >18
* History of cancer diagnosis, previously treated with at least 8 infusions of chemotherapy regimen that included oxaliplatin or at least 6 infusions of chemotherapy regimen that included cisplatin, paclitaxel, docetaxel, or any combination of these.
* No ongoing pain in distal symmetric distribution (subjects with symptoms and signs such as mild numbness, or vibration sensation loss are eligible to be included in the control group).
* Able and willing to sign an IRB-approved written informed consent. * Subjects in the control group will be matched by the type of previous chemotherapy to the subjects in the Painful CIPN group. An additional attempt will be made to match controls by sex, age, cancer diagnosis, and cumulative neurotoxic chemotherapy dose.

Exclusion Criteria:

* History of pre-existing painful distal symmetric polyneuropathy prior to chemotherapy.
* Alternative etiology exists for the distal painful symptoms.
* Current or previous treatment with a vinca alkaloid (e.g. vincristine, vinblastine), bortezomib, or another agent which may cause major peripheral neurotoxicity.
* Pregnant
* Concomitant medication as follows:
* Patients receiving chronic daily opioids, topical lidocaine or topical capsaicin will be excluded.
* Patients receiving as needed (PRN) analgesics, including acetaminophen, NSAIDs or short-acting opioids, will be required not to take them 48h before testing, at for at least five half-lives of the specific analgesic, at the discretion of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Haroutounian, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the recent proposal from the International Committee of Medical Journal Editors, patient-level data will be made available within 6 months after publication of the primary manuscript. Data will be provided to researchers who submit a methodologically sound research proposal including a protocol and statistical analysis plan. No patient-identifying fields (including dates) will be included in the shared dataset. Certain technical data related to the intellectual property rights of LasMed LLC may not be available for sharing.
Supporting Information: Study Protocol, ICF
Time Frame: Patient-level data will be made available within 6 months after publication of the primary manuscript.
Access Criteria: Data will be provided to researchers who submit a methodologically sound research proposal including a protocol and statistical analysis plan. No patient-identifying fields (including dates) will be included in the shared dataset. Certain technical data related to the intellectual property rights of LasMed LLC may not be available for sharing.

REFERENCES:
- [Derived] Nemenov MI, Alaverdyan H, Burk C, Roles K, Frey K, Yan Y, Kazinets G, Haroutounian S. Characterization of Patients With and Without Painful Peripheral Neuropathy After Receiving Neurotoxic Chemotherapy: Traditional Quantitative Sensory Testing vs C-Fiber and Adelta-Fiber Selective Diode Laser Stimulation. J Pain. 2022 May;23(5):796-809. doi: 10.1016/j.jpain.2021.11.011. Epub 2021 Dec 9. PMID 34896646
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at Washington University in St Louis School of Medicine. Participants were recruited between September 17, 2018, and September 17, 2019.
Pre-assignment Details: This is a case-control study. Case group: Patients with current symptoms of painful chemotherapy-induced peripheral neuropathy (CIPN) following treatment with oxaliplatin, cisplatin, paclitaxel, or docetaxel. Control group: patients who received the same chemotherapy agents, but who did not report current (or other long-term) painful CIPN.
Groups:
- Group A: Painful Neuropathy Group: Patient with painful neuropathy after receiving treatment with oxaliplatin, cisplatin, paclitaxel or docetaxel
- Group B: Control Group: Patient with no painful CIPN after receiving treatment with ...
Period: Overall Study
Arm/Group | Group A: Painful Neuropathy Group | Group B: Control Group
Started | 22 | 20
Completed | 20 | 20
Not Completed | 2 | 0
Not completed — visit scheduling conflicts | 2 | 0

BASELINE CHARACTERISTICS:
Population: Since this is a case-control study only patients completed the study visit are reported here.
Groups:
- Group A: Painful CIPN Group: Patients after chemotherapy with painful neuropathy
- Group B: Control Group: Patients after chemotherapy without painful neuropathy
- Total: Total of all reporting groups
Arm/Group | Group A: Painful CIPN Group | Group B: Control Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 17 | 31
  >=65 years | 6 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (10.6) | 50.5 (14.5) | 54.3 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 17 | 19 | 36
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Aδ:C Fiber Detection Threshold Ratio
Description: Comparison of the Aδ:C fiber detection threshold ratio (as measured by the DLss) between patients with painful neuropathy and patients who did not develop painful neuropathy following similar cancer chemotherapy
Time Frame: At the time of the DLss (day 1)
Population: Enrolled patients from control and case groups who completed Aδ:C fiber detection threshold ratio testing by DLss
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Group A: Painful Neuropathy Group: -patients after chemotherapy with painful CIPN who completed Aδ:C fiber detection threshold ratio testing by DLss.
- Group B: Control Group: -patients after chemotherapy who did not report current (or other long-term) painful CIPN and completed Aδ:C fiber detection threshold ratio testing by DLss.
Arm/Group | Group A: Painful Neuropathy Group | Group B: Control Group
Number analyzed (Participants) | 20 | 19
ratio | 2.04 (0.74) | 1.57 (0.39)
Statistical Analysis 1: Comparison: Group A: Painful Neuropathy Group vs Group B: Control Group; Test type: Other — Multivariable logistic regression was applied to predict binary outcome while controlling for other potential confounding factors (age, cumulative chemotherapy dose, chemotherapy group); p = 0.05, Regression, Logistic — threshold for p value is 0.05; Slope = -0.130

2. Secondary Outcome: The Aδ:C Pain Threshold Ratio
Description: Aδ:C pain threshold shows Aδ fiber threshold divided by C fiber threshold measured by DLss detection and pain threshold protocols.
Time Frame: At the time of the DLss (day 1)
Population: Aδ:C threshold ratios were measured among patients from both groups. Only patients who finished DLss testing for pain threshold determination were included in analysis.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group A: Painful Neuropathy Group | Group B: Control Group
Number analyzed (Participants) | 18 | 16
ratio | 1.95 (0.71) | 1.60 (0.42)
Statistical Analysis 1: Comparison: Group A: Painful Neuropathy Group; Test type: Other — Spearman correlation coefficient between the Aδ:C fiber detection threshold ratio and the severity of painful CIPN on NPSI scale for patients with painful CIPN was calculated; p = 0.7525, Spearman's correlation coefficient — The thrshold for p value is 0.05; rho coefficient = 0.22
Statistical Analysis 2: Comparison: Group B: Control Group; Test type: Other — Spearman correlation coefficient between the Aδ:C fiber detection threshold ratio and the severity of painful CIPN on NPSI scale for Control group patients without painful CIPN was calculated; p = 0.1876, Spearman's correlation coefficien — The threshold for p value is 0.05; rho coefficient = 0.32
Statistical Analysis 3: Comparison: Group A: Painful Neuropathy Group; Test type: Other — Spearman correlation coefficient between the Aδ:C fiber pain threshold ratio and the severity of painful CIPN on NPSI scale for patients with painful CIPN was calculated; p = 0.61, Spearman's correlation coefficient — The threshold for p value is 0.05; rho coefficient = 0.13
Statistical Analysis 4: Comparison: Group B: Control Group; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.2914, Spearman's correlation coefficient — The threshold for p value is 0.05; rho coefficient = -0.2812205

3. Secondary Outcome: The Severity of Neuropathy on NPSI Scale.
Description: The severity of painful CIPN on Neuropathic Pain Symptom Inventory (NPSI) scale.
  Increased NPSI (0-100) score indicates more severe neuropathic pain.
Time Frame: At the time of the DLss (day 1)
Population: Only patients who completed NPSI questionnaire were included in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Group A: Painful Neuropathy Group: -patients after chemotherapy with painful CIPN who completed NPSI questionnaire were included in the analysis.
- Group B: Control Group: -patients after chemotherapy who did not report current (or other long-term) painful CIPN and completed NPSI questionnaire were included in the analysis.
Arm/Group | Group A: Painful Neuropathy Group | Group B: Control Group
Number analyzed (Participants) | 20 | 20
score on a scale | 32.60 (19.89) | 0.2 (0.7)

ADVERSE EVENTS:
Time Frame: Since study activities included relatively safe testings conducted within a day the safety data were actively collected during study visit day. Patients were informed to report any adverse effects throughout the study visit day, and by telephone any time after the study visit.
Description: any unfavorable medical occurrence in a human subject including any abnormal sign, symptom, or disease.
Groups:
- Group A: Painful CIPN Group: All patients who were enrolled in the Case group and completed any testing
- Group B: Control Group: All patients who were enrolled in the Control group and completed any testing
Arm/Group | Group A: Painful CIPN Group | Group B: Control Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Painful CIPN Group (N=20) | Group B: Control Group (N=20)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — increased sensitivity and pain in the right foot after testing. Duration: 30 minutes. Self-resolved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT03687970/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-02): https://cdn.clinicaltrials.gov/large-docs/70/NCT03687970/ICF_001.pdf